CLINICAL TRIAL: NCT02279615
Title: EFFICACY AND SAFETY OF COMBINATION THERAPY WITH β3-ADRENOCEPTOR AGONIST (MIRABEGRON) AND α-ADRENOCEPTOR ANTAGONIST (TAMSULOSIN) FOR TREATMENT OF OVERACTIVE BLADDER IN MALE PATIENTS WITH BENIGN PROSTATIC HYPERPLASIA.
Brief Title: Efficacy And Safety Of Combination Therapy For Treatment Of Overactive Bladder In Male Patients With Benign Prostatic Hyperplasia.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MIRTAM-2014OB
Record Dates: First submitted 2014-10-10; First posted 2014-10-31 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Overactive Bladder; Benign Prostatic Hyperplasia
Keywords: Overactive Bladder; Benign Prostatic Hyperplasia; Combination Therapy; β3-Adrenoceptor Agonist; Mirabegron; Myrbetriq; α-Adrenoceptor Antagonist; Tamsulosin; Flomax
MeSH Terms: conditions — Urinary Bladder, Overactive; Prostatic Hyperplasia | interventions — mirabegron; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): (Mirabegron + Tamsulosin)
  Interventions: Drug: Mirabegron; Drug: Tamsulosin
- Control Group (Placebo Comparator): (Placebo + Tamsulosin)
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Mirabegron — 50mg of mirabegron per day will be given.
  Other Names: Myrbetriq
  Arms: Treatment Group
Drug: Tamsulosin — 0.4mg of flomax per day.
  Other Names: Flomax

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of combination therapy involving β3-adrenoceptor agonist, mirabegron, and α-blockers for the treatment of OAB symptoms in male patients with BPH.

DETAILED DESCRIPTION:
Mirabegron (MyrbetriqTM, Astellas Pharma Inc.) is a drug that is approved by the FDA for the treatment of overactive bladder (OAB) with symptoms of urinary frequency, urgency and urgency incontinence. Multiple studies have shown that this drug also has the potential to improve patient tolerability, compliance and subsequent patient quality of life without inducing unfavourable adverse events commonly associated with antimuscarinic medications. These adverse events include, but are not limited to, dry mouth, constipation, confusion, and acute urinary retention (AUR).

Studies now have shown that mirabegron may also provide an effective treatment option for OAB in men with benign prostatic hyperplasia (BPH) without inducing the above mentioned adverse events. This study will look at the combination therapy of Mirabegron and Tamsulosin, versus Tamsulosin and placebo alone to prove that this treatment (Mirabegron and Tamsulosin) is effective for those men who suffer from both overactive bladder along with benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Male patients over the age of 50
* Clinical BPH on stable dose of alpha-blocker therapy for more than 1 month
* OAB symptoms (frequency, urgency, nocturia, urgency incontinence)

Exclusion Criteria:

* Post-void residual (PVR) > 200mL
* Active, culture-proven urinary tract infection
* Acute/chronic prostatitis
* Previous lower urinary tract malignancy (i.e. bladder, prostate malignancy)
* History of cystolithiasis
* Previous pelvic surgery (i.e. prostatectomy, cystectomy, recent pelvic/endourologic instrumentation including cystoscopy, nephroscopy, ureteral stent insertion, Transrectal Ultrasound (TRUS) biopsy)
* Previous pelvic radiation

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | Treatment period: 4 weeks
  Measured before and after combination therapy.
Quality of Life Score (QoLS) | Treatment period: 4 weeks
  Measured before and after combination therapy
Overactive Bladder Symptom Score (OABSS) | Treatment period: 4 weeks
  Measured before and after combination therapy

SECONDARY OUTCOMES:
Adverse Events | Timeline: 4 weeks
  Measured during treatment of combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton - McMaster Institute of Urology, Hamilton, Ontario, Canada